CLINICAL TRIAL: NCT04343729
Title: Efficacy of Injectable Methylprednisolone Sodium Succinate in the Treatment of Patients With Signs of Severe Acute Respiratory Syndrome Under the New Coronavirus (SARS-CoV2): a Phase IIb, Randomized, Double-blind, Placebo-controlled, Clinical Trial.
Brief Title: Methylprednisolone in the Treatment of Patients With Signs of Severe Acute Respiratory Syndrome in Covid-19
Acronym: MetCOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAEE: 30615920.2.0000.0005
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: SARS-CoV Infection; Severe Acute Respiratory Syndrome (SARS) Pneumonia
Keywords: SARS-CoV-2; Covid-19; Corticosteroid; Severe Acute Respiratory Syndrome (SARS) Pneumonia; Coronavirus; methylprednisolone
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Pneumonia; COVID-19; Coronavirus Infections | interventions — Methylprednisolone Hemisuccinate; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone (Active Comparator): 0.5mg/kg injectable methylprednisolone sodium succinate, twice daily, for 5 days.
  Interventions: Drug: Methylprednisolone Sodium Succinate
- Placebo (Placebo Comparator): Saline solution, twice daily, for 5 days. Injectable.
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: Methylprednisolone Sodium Succinate — injectable solution at a dose of 0.5mg/kg
  Other Names: methylprednisolone
  Arms: Methylprednisolone
Drug: Placebo solution — injectable saline solution
  Other Names: placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, phase IIb clinical trial to assess the efficacy of injectable methylprednisolone sodium succinate (MP) in patients with severe acute respiratory syndrome (SARS) in COVID-19 infection. A total of 416 individuals of both sexes, aged over 18 years old, with symptoms suggestive or confirmed diagnosis of severe acute respiratory syndrome (SARS), hospitalized at the Hospital and Pronto-Socorro Delphina Rinaldi Abdel Aziz (HPSDRAA), with clinical and radiological findings suggestive of SARS-CoV2 infection, will be randomized at a 1:1 ration to receive either MP (0.5mg/kg of weight, twice daily, for 5 days) or placebo (saline solution, twice daily, for 5 days).

ELIGIBILITY:
Inclusion Criteria:

1. Suspected cases of COVID-19, from clinical and radiological data, during the pandemic;
2. Adult aged 18 years or older, at the time of inclusion (children under 18 will not be included due to the recognized lower lethality in previous published studies, and the difficulty of consent in the context of an emergency in public health);
3. SpO2 ≤ 94% in room air OR in use supplementary oxygen OR under invasive mechanical ventilation

Exclusion Criteria:

1. History of hypersensitivity to MPS;
2. People living with HIV and AIDS;
3. Chronic use of corticosteroids or immunosuppressive agents;
4. Pregnancy or breastfeeding;
5. Decompensated cirrhosis;
6. Chronic renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2020-04-18 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Mortality rate at day 28 | on day 28, after randomization
  Mortality rate on day 28, after randomization

SECONDARY OUTCOMES:
Mortality rate on days 7, 14 and 28 | after randomization, up to 28 days.
  Proportion of patient that died on days 7, 14 and 28.
Incidence of orotracheal intubation | after randomization, up to 7 days.
  proportion of patients requiring orotracheal intubation
Change in oxygenation index | after randomization, up to 7 days.
  Proportion of patients with oxygenation index (PaO2 / FiO2) < 100 in 7 days.

OTHER OUTCOMES:
Spirometry (exploratory outcome) | 120 days after randomization
  Forced expiratory capacity at the first second of exhalation (FEV1) in liters
Spirometry (exploratory outcome) | 120 days after randomization
  Forced vital capacity (FVC) in liters
Spirometry (exploratory outcome) | 120 days after randomization
  FEV1/FVC ratio
Spirometry (exploratory outcome) | 120 days after randomization
  Forced expiratory flow (FEF) in cmH2O
Spirometry (exploratory outcome) | 120 days after randomization
  Peak expiratory flow (PEF) in cmH2O

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital e Pronto Socorro Delphina Rinaldi Abdel Aziz, Manaus, Amazonas, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all patient data will be shared after study publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after study publication.
Access Criteria: upon formal request.

REFERENCES:
- [Derived] Barros CMSS, Freire RS, Frota E, Rezende Santos AG, Farias MEL, Rodrigues MGA, Silva BM, Prado Jeronimo CM, Netto RLA, Silva Borba MG, Baia-da-Silva D, Brito-Sousa JD, Xavier MS, Araujo-Alexandre MA, Sampaio VS, Melo GC, Areas GT, Hajjar LA, Monteiro WM, Gomes Naveca F, Costa FTM, Val FFA, Lacerda MVG; Metcovid team. Short-Course of Methylprednisolone Improves Respiratory Functional Parameters After 120 Days in Hospitalized COVID-19 Patients (Metcovid Trial): A Randomized Clinical Trial. Front Med (Lausanne). 2021 Nov 30;8:758405. doi: 10.3389/fmed.2021.758405. eCollection 2021. PMID 34917633
- [Derived] Jeronimo CMP, Farias MEL, Val FFA, Sampaio VS, Alexandre MAA, Melo GC, Safe IP, Borba MGS, Netto RLA, Maciel ABS, Neto JRS, Oliveira LB, Figueiredo EFG, Oliveira Dinelly KM, de Almeida Rodrigues MG, Brito M, Mourao MPG, Pivoto Joao GA, Hajjar LA, Bassat Q, Romero GAS, Naveca FG, Vasconcelos HL, de Araujo Tavares M, Brito-Sousa JD, Costa FTM, Nogueira ML, Baia-da-Silva DC, Xavier MS, Monteiro WM, Lacerda MVG; Metcovid Team. Methylprednisolone as Adjunctive Therapy for Patients Hospitalized With Coronavirus Disease 2019 (COVID-19; Metcovid): A Randomized, Double-blind, Phase IIb, Placebo-controlled Trial. Clin Infect Dis. 2021 May 4;72(9):e373-e381. doi: 10.1093/cid/ciaa1177. PMID 32785710